CLINICAL TRIAL: NCT05781386
Title: An Open-label, Phase I Trial of SIM1811-03 to Assess the Safety, Efficacy and Pharmacokinetics/Pharmacodynamics in Subjects With Advanced Tumors
Brief Title: A Phase I Trial of SIM1811-03 in Subjects With Advanced Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Biologics Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM1811-03-TNFR2-101
Record Dates: First submitted 2023-01-31; First posted 2023-03-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor; Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIM1811-03 monotherapy or SIM1811-03 in combination with Sintilimab injection (Experimental): All participants receive SIM1811-03 or SIM1811-03 in combination with Sintilimab injection
  Interventions: Drug: SIM1811-03 or in combination with Sintilimab injectiont

INTERVENTIONS:
Drug: SIM1811-03 or in combination with Sintilimab injectiont — SIM1811-03 is a first-in-class igG-1 based humanized anti-tumor necrosis factor type 2 receptor (TNFR2) monoclonal antibody for the treatment of malignant tumor.
  Sintilimab is an IgG4 humanized monoclonal antibody against programmed cell death protein 1 (PD-1)

SUMMARY:
This is a first in human, open-label, dose escalation and expansion Phase I study of SIM1811-03 in adult patients with advanced tumors. SIM1811-03 is a first-in-class IgG1-based humanized anti-tumor necrosis factor type 2 receptor (TNFR2) monoclonal antibody for the treatment of malignant tumors.

DETAILED DESCRIPTION:
This is a phase I trial to evaluate the safety, efficacy, and pharmacokinetic/ pharmacodynamic characteristics of SIM1811-03 in participants with advanced tumors.

The trial is composed of two parts, Part I and Part II. Part I is a dose escalation part to determine the MTD and/or RD of SIM1811-03 or SIM1811-03 in combination with Sintilimab Injection . Part II is a dose expansion part at RD level SIM1811-03 determined in Part I to assess the anti-tumor activity of SIM1811-03 or SIM1811-03 in combination with Sintilimab Injection in participants with advanced solid tumors or CTCL. The tumor types in Part II will be adjusted based on the response observed in Part I.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent must be obtained prior to any procedures that are not considered standard of care.
2. ≥18 years old on the day of signing informed consent, male or female;
3. Histologically and/or cytologically documented advanced/metastatic solid tumors or histologically confirmed CTCL;
4. Have relapsed or refractory advanced solid tumors or CTCL, whose disease has progressed during or after standard therapy
5. At least one measurable tumor lesion (RECIST 1.1) for participants with solid tumors. Tumor lesions previously treated with radiotherapy or local therapy should not be considered as measurable unless progression is documented.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
7. Life expectancy of ≥ 12 weeks.
8. Adequate organ and marrow functions 9） Provide archived or fresh biopsy tumor tissue samples or tissue sections

10) Females of childbearing potential require strict contraception during the study.

Exclusion Criteria:

1) Participated in an interventional clinical trial or has used investigational devices within 28 days prior to first dose of study drug or received systemic anti-cancer treatments.

2）Toxicity due to previous antineoplastic therapy has not recovered to grade 0 or 1 unless such AEs are not considered to pose safety risks.

3) Required use of corticosteroids for more than 7 consecutive days within 14 days prior to the first dose of study treatment.

4) Participated with active or history of or risk of autoimmune disease 5) Major surgery (except biopsy) or unhealed wound within 4 weeks prior to first dose of study drug.

6) Other known malignancies within 2 years prior to enrollment. 7) Has known active central nervous system (CNS) metastases. 8) History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, symptomatic interstitial lung disease or evidence of active pneumonia that is not considered appropriate by the investigator.

9) Participants with a history of active pulmonary tuberculosis infection within 1 year prior to first dose of study drug.

10) History of hemorrhagic disease requiring transfusion within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-03-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Part I The maximum tolerated dose (MTD) or recommended dose (RD) | Within 28 days after the first dose in Q2W; Within 21 days after the first dose in Q3W
  Part I (dose escalation): To estimate the maximum tolerated dose (MTD) or recommended dose (RD) of SIM1811-03 Monotherapy or in combination with sintilimab
Part II ORR for Solid Tumor | Q2W: Participants will be evaluated every 8 weeks from baseline to Treatment Cycle 12 (an average of 1 year); Q3W:Participants will be evaluated every 6 weeks from baseline to Treatment Cycle 12 (an average of 1 year)
  Solid tumors: objective response rate (ORR) assessed by Investigator per RECIST 1.1 from baseline to disease progression
Part II ORR for CTCL | Q2W:Participants will be evaluated every 8 weeks from baseline to Treatment Cycle 12 (an average of 1 year); Q3W:Participants will be evaluated every 6 weeks from baseline to Treatment Cycle 12 (an average of 1 year)
  CTCL: ORR assessed by Investigator per global response score

SECONDARY OUTCOMES:
safety and tolerability (incidence of AE and SAE) | All AEs/SAEs will be collected in this study from the time the subject signs the informed consent form until 90 days after the last dose
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | from Cycle 1 to Last dose (an average of 1 year)
  Serum concentrations of study drugs
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | from Cycle 1 to Last dose (an average of 1 year)
  Area under the concentration-time curve (AUC)
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | from Cycle 1 to Last dose (an average of 1 year)
  Maximum concentration (Cmax)
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | from Cycle 1 to Last dose (an average of 1 year)
  Pre-dose (trough) concentration (Ctrough)
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | from Cycle 1 to Last dose (an average of 1 year)
  Time to maximum concentration (Tmax)
Pharmacokinetics profile of SIM1811-03 and in combination with Sintilimab | Collection point would Predose, 0 hour, 24 hours, 168hours, 336 hours post-dose from Cycle 1 to Last dose (an average of 1 year)
  Half-life (T1/2)
Antidrug antibodies of SIM1811-03 and Sintilimab | before staring the treatment for the first 7 treatment cycles (each cycle would be 28 days/21 days)
  Incidence of serum antidrug antibodies.
Neutralizing antibodies of SIM1811-03 and Sintilimab | before staring the treatment for the first 7 treatment cycles (each cycle would be 28 days/21 days)
  Incidence of neutralizing antibodies to study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao Z, Zhang Q, Chen H, Chen J, Kang J, Yu H, Song Y, Zhang X. TNFR2 promotes pancreatic cancer proliferation, migration, and invasion via the NF-kappaB signaling pathway. Aging (Albany NY). 2023 Aug 16;15(16):8013-8025. doi: 10.18632/aging.204941. Epub 2023 Aug 16. PMID 37589506